CLINICAL TRIAL: NCT04475653
Title: Benefit of Wearing an Activity Tracker in Sarcoidosis
Acronym: ildfitbit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ild care foundation (Other); St. Antonius Hospital (Other); Gelderse Vallei Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ildcarefitbit2017
Record Dates: First submitted 2020-07-01; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Sarcoidosis; Fatigue
Keywords: Physical Activity; Exercise Capacity; Activity Tracker
MeSH Terms: conditions — Sarcoidosis; Fatigue; Motor Activity

STUDY DESIGN:
Intervention Model Description: This prospective, randomized clinical trial included 54 sarcoidosis patients who received an AT (Group Ia: 27 with coaching and Group Ib: 27 without). Exercise capacity and fatigue scores (Fatigue Assessment Scale) were evaluated at baseline and after three months. A historical group of sarcoidosis patients (Group II; n=41) from an earlier study who did not follow a physical activity program served as controls.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group coaching (Active Comparator): Performing physical activities with Activity tracker, coaching included
  Interventions: Behavioral: Physical Activity using an Activity Tracker
- Group Independant (Active Comparator): Performing physical activities with Activity tracker, coaching NOT included
  Interventions: Behavioral: Physical Activity using an Activity Tracker
- Controls (Other): Controls from former study (see Study description)
  Interventions: Behavioral: Physical Activity using an Activity Tracker

INTERVENTIONS:
Behavioral: Physical Activity using an Activity Tracker

SUMMARY:
Sarcoidosis causes many disabling symptoms, including fatigue, muscle weakness, and exercise limitations. Physical activity programs have been shown to improve physical performance and decrease fatigue in sarcoidosis.

Objectives: The aim of this study was to evaluate (1) the effect of continuous activity monitoring using an electronic activity tracker (AT), compared to controls, and (2) the effect of additional personal coaching on exercise performance and fatigue of sarcoidosis patients.

Method: This prospective, randomized clinical trial included 54 sarcoidosis patients who received an AT (Group Ia: 27 with coaching and Group Ib: 27 without). Exercise capacity and fatigue scores (Fatigue Assessment Scale) were evaluated at baseline and after three months. A historical group of sarcoidosis patients (Group II; n=41) from an earlier study who did not follow a physical activity program served as controls.

DETAILED DESCRIPTION:
Sarcoidosis patients often suffer not only from organ-related symptoms but also from disabling non-specific, non-organ-related symptoms, such as fatigue, reduced muscle strength, loss of physical condition, reduction of physical activity (PA) in daily life and pain. Fatigue is the most frequently reported in sarcoidosis patients disregarding the clinical presentation, varying from 50 to 90%. This may persist after other signs of sarcoidosis activity have resolved, and adversely impacts major life areas, including quality of life (QoL) and work ability.

So far, there is promising evidence for the benefits of physical training in sarcoidosis. Interventions involving technology that is readily accessible on a daily basis to monitor activity levels can support care providers in encouraging patients to achieve behavioral changes. These interventions may be an effective strategy to provide PA-coaching without increasing time demands on primary care providers. Moreover, they give patients an opportunity to keep up a more active lifestyle with direct feedback and monitor their physical performance over time. Counseling, guidance and support using e-health technology had been found to be very helpful for patients who want to improve their PA. The use of commercially available, technology-based wearable activity trackers (ATs) such as Fitbit is growing for research and recreational purposes, both among healthy persons and among those with chronic illness. Beneficial effects of AT-based counseling have been demonstrated in patients with chronic diseases. In a recent study by our group we found that wearing an AT stimulated patients to be more physically active.

The aim of this study was to evaluate (1) the effect of continuous activity monitoring using an electronical AT and (2) the effect of additional personal coaching of sarcoidosis patients. The outcome measures were exercise performance and fatigue.

Intervention All participants received a Fitbit for free. They were encouraged to improve their physical fitness, which was assessed at baseline. The patients in the intervention group (group Ia) engaged in a three-month physical therapist-guided activity program. The guidance was based on the input from the AT and the questionnaires. The weekly FAS scores, Fitbit-measured parameters and brief daily questions were combined in a web-based dashboard accessible to the assigned physical therapist. The information was used for goal setting, encouraging, and identifying barriers and facilitators for patients becoming more active. The coaching procedure included weekly action planning and feedback, modelling of behaviors and problem solving, and individual decision making by email and/or telephone. The coaching physical therapist acted as facilitator, and assisted participants in making choices and achieving success in terms of reaching self-selected goals.

Although the patients in group Ib did not receive the guidance from a physical therapist, their daily activity was also computed with the Fitbit Charge HR (Brand name), and patients were also able to use a Fitbit and monitor app to monitor their performance, questionnaire results and progress.

Self-report feedback questionnaires at follow-up (12 weeks) were used to determine participants' experience with data from the Fitbit tracker itself and coaching, if applicable.

ELIGIBILITY:
Inclusion Criteria:

* participants being in a clinically stable condition
* no change in initiated medical management during the preceding three months
* having sufficient command of the Dutch language
* having internet access at home or a compatible smartphone/tablet.

Exclusion Criteria:

- Patients participated in a training program during the six months prior to inclusion were excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-07-08 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
6 Minute Walking Distance (MWD) | 3 months
  Change from baseline in 6 MWD in 3 months
Fatigue monitoring | 3 months
  Fatigue was measured with the 10-item Fatigue Assessment Scale (FAS) [9]. This questionnaire was filled out on a weekly basis. Outcome measure: Change from baseline in fatigue during 3 months.
  FAS scores 10 - 21: no fatigue (normal) FAS scores 22 - 50: substantial fatigue
  Subscores:
  * fatigue: scores 22-34
  * extreme fatigue: scores ≥ 35
  The Minimal Important Difference (MCID) is at least 4 points or 10% change of the baseline value.
Steep ramp test (SRT) | 3 months
  Exercise performance protocol on a cycle ergometer. Outcome: Change from baseline and after 3 months intervention of physical activity

SECONDARY OUTCOMES:
Lung function tests | 3 months
  Forced vital capacity (FVC) and forced expiratory volume in one second (FEV1) were measured with a pneumotachograph. The diffusing capacity of the lung for carbon monoxide (DLCO) was measured using the single-breath method (Masterlab, Jaeger, Würzburg, Germany). Values were expressed as a percentage of the predicted value (i.e., FVC%, FEV1%, and DLCO% respectively).
  Outcome measure: Change baseline and after 3 months intervention

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein Drent, MD, PhD, Study Chair — ild care foundation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.ildcare.nl/index.php/benefits-of-e-health-based-coaching-of-physical-training-in-patients-with-ild/